CLINICAL TRIAL: NCT03699241
Title: A Randomized, Double-blinded, Placebo-controlled, Dose-escalation Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant HIV Envelope Protein BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, in Healthy, HIV-1 Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: GlaxoSmithKline (Industry); Fred Hutchinson Cancer Research Center - Seattle HIV Vaccine Trials Unit (Unknown); Kenya AIDS Vaccine Initiative - Institute of Clinical Research (KAVI-ICR) (Unknown); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAVI W001
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Placebo Comparator): HIV-Uninfected participants
  Interventions: Biological: BG505 SOSIP.664 gp140, adjuvanted; Biological: Placebo
- Group 2 (Placebo Comparator): HIV-Uninfected participants
  Interventions: Biological: BG505 SOSIP.664 gp140, adjuvanted; Biological: Placebo
- Group 3 (Placebo Comparator): HIV-Uninfected participants
  Interventions: Biological: BG505 SOSIP.664 gp140, adjuvanted; Biological: Placebo
- Group 4 (Placebo Comparator): HIV-Uninfected participants
  Interventions: Biological: BG505 SOSIP.664 gp140, adjuvanted; Biological: Placebo
- Group 5 (Placebo Comparator): HIV-Uninfected participants
  Interventions: Biological: BG505 SOSIP.664 gp140, adjuvanted; Biological: Placebo

INTERVENTIONS:
Biological: BG505 SOSIP.664 gp140, adjuvanted — Dosage of 30ug, Intramuscular administration
  Arms: Group 1; Group 4
Biological: BG505 SOSIP.664 gp140, adjuvanted — Dosage of 100ug, Intramuscular administration
  Arms: Group 2; Group 5
Biological: BG505 SOSIP.664 gp140, adjuvanted — Dosage of 300ug, Intramuscular administration
  Arms: Group 3
Biological: Placebo — Tris-NaCl Diluent

SUMMARY:
This a phase 1 first-in-human clinical trial to evaluate the safety, tolerability, and immunogenicity of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, in up to 60 healthy adult HIV-uninfected volunteers.

DETAILED DESCRIPTION:
This a phase 1 first-in-human clinical trial to evaluate the safety, tolerability, and immunogenicity of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, in up to 60 healthy adult HIV-uninfected volunteers. BG505 SOSIP.664 gp140 is a stable, soluble, cleaved HIV envelope trimer formulated in 0.55mL at 2mg/mL in 20 mM Tris, 100 mM NaCl, pH 7.5 and will be administered IM.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female, including transgender individuals, as assessed by a medical history, physical exam, and laboratory tests
2. At least 18 years of age on the day of screening and has not reached his/her 51st birthday on the day of first vaccination
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study
4. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and potential impact and/or risks linked to vaccination and participation in the trial; written informed consent will be obtained from the volunteer before any study-related procedures are performed
5. Willing to undergo HIV testing, risk reduction counselling and receive HIV test results
6. All volunteers born female engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception for 4 months following investigational product administration
7. All volunteers born female, who are not heterosexually active at screening, must agree to utilize an effective method of contraception if they become heterosexually active
8. All volunteers born female must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Procedures (Appendix A and B)
9. All sexually active volunteers born male, regardless of reproductive potential, must be willing to use an effective method of contraception (such as consistent condom use) from the day of first vaccination until at least 4 months after the last vaccination to avoid exposure of partners to investigational product in ejaculate and to prevent conception with female partners
10. Willing to forgo donations of blood, or any other tissues during the study and, for those who test HIV-positive due to vaccine-induced antibodies, until the anti-HIV antibody titers become undetectable

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of corticosteroids (the use of topical, nasal, or inhaled steroids is permitted), immunosuppressive, anticancer, anti-tuberculosis or other medications considered significant by the investigator within the previous 6 months. The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 2 weeks prior to enrolment in this study
3. Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the investigator makes the volunteer unsuitable for participation in the study
4. Reported risky behavior for HIV infection within 12 months prior to vaccination
5. If female, pregnant or planning a pregnancy during the period of enrolment until 4 months after the last study vaccination; or lactating
6. Bleeding disorder that was diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions.) (Note: A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has IM injections and blood draws without any adverse experience, is eligible)
7. Infectious disease: chronic hepatitis B infection (HbsAg-positive), current hepatitis C infection (for US sites: HCV Ab positive and HCV RNA positive, for African site: HCV Ab positive only) treatment for chronic hepatitis C infection in the past year, or active syphilis (positive RPR confirmed by TPHA); active tuberculosis (for African site only)
8. History of splenectomy
9. Any of the following abnormal laboratory parameters listed below:

   Hematology
   * Absolute Neutrophil Count (ANC) - all volunteers: ≤1,000/mm3
   * Absolute Lymphocyte Count (ALC) - all volunteers: ≤650/mm3
   * Hemoglobin - African volunteers: <9.5 g/dl in females; <11.0 g/dl in males
   * Hemoglobin - US volunteers: <10.5 g/dl in females; <11.0 g/dl in males
   * Platelets - African volunteers: <100,000 cells/mm3
   * Platelets - US volunteers: <125,000 cells/mm3

   Chemistry
   * Creatinine >1.1 x upper limit of normal (ULN)
   * ALT >1.25 x ULN
   * AST >1.25 x ULN

   Urinalysis

   Clinically significant abnormal dipstick confirmed by microscopy:
   * Protein = 1+ or more
   * Blood = 2+ or more (not due to menses)
10. Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after vaccination with Investigational Product; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product. (Exception is live attenuated influenza vaccine within 14 days)
11. Receipt of blood transfusion or blood-derived products within the previous 3 months
12. Participation in another clinical trial of an Investigational Product currently, within the previous 3 months or expected participation during this study; Concurrent participation in an observational study not requiring any blood or tissue sample collection is not an exclusion
13. Prior receipt of another investigational HIV vaccine candidate or HIV monoclonal antibody (Note: receipt of placebo in a previous HIV vaccine trial will not exclude a volunteer from participation if documentation is available and the Medical Monitor gives approval)
14. History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration)
15. Psychiatric condition that compromises safety of the volunteer and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years prior to screening, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
16. Seizure disorder: A participant who has had a seizure in the last 3 years prior to screening is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years)
17. A history of malignancy in the past 5 years (prior to screening) or ongoing malignancy (A history of a completely excised malignancy that is considered cured is not an exclusion)
18. Active, serious infections requiring parenteral antibiotic, antiviral or antifungal therapy within 30 days prior to enrolment
19. Body mass index (BMI) ≥35
20. Body weight <110 pounds (55 kg); for US sites only
21. If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers with moderate or greater reactogenicity (i.e., solicited adverse events) during a 7-day follow-up period after each vaccination | 7 days post-vaccination
  To evaluate the safety and tolerability of the study regimens based on the frequency of local and systemic reactogenicity events as assessed using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (v2.1).
Proportion of volunteers with moderate or greater and/or vaccine related unsolicited adverse events (AEs), including safety laboratory (biochemical, haematological) parameters, from the day of each vaccination up to 28 days post each vaccination | 28 days post-vaccination
  To evaluate the safety and tolerability of the study regimens based on the proportion of volunteers with moderate or greater unsolicited adverse events including safety laboratory as assessed using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (v2.1).
Proportion of volunteers with vaccine-related serious adverse events (SAEs) throughout the study period | 18 months
  To evaluate the safety and tolerability of the study regimens based on the proportion of volunteers with vaccine-related serious adverse events including safety laboratory as assessed using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (v2.1).
Proportion of volunteers in each group with potential immune-mediated diseases (pIMD) from the day of injection throughout the study period | 18 months
  To evaluate the proportion of volunteers in each group with potential immune-mediated diseases (pIMDs) based on a defined list of pIMDs in the study protocol.

SECONDARY OUTCOMES:
To assess immune responses elicited by the different BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, doses: | 20 months
  Proportion of volunteers with neutralizing antibodies against autologous BG505 SOSIP.664 gp140 Vaccine, Adjuvanted
To assess immune responses elicited by the different BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, doses: | 20 months
  Proportion of volunteers with and magnitude of trimer binding antibodies to BG505 SOSIP.664 gp140 Vaccine, Adjuvanted
To assess immune responses elicited by the different BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, doses: | 20 months
  Proportion of volunteers with neutralizing antibodies against additional viral strains (e.g., Tier 1a/b, Tier 2)
To assess immune responses elicited by the different BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, doses: | 20 months
  Proportion of volunteers with and magnitude of binding antibodies to HIV Env
To assess immune responses elicited by the different BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, doses: | 20 months
  Proportion of volunteers with HIV Env specific B and T-cell responses

CONTACTS AND LOCATIONS:
Overall Officials: Julie McElrath, MD, PhD, Principal Investigator — Seattle HIV Vaccine Trials Unit; Omu Anzala, MBChB, PhD, Principal Investigator — Kenya AIDS Vaccine Initiative - Institute of Clinical Research (KAVI-ICR); Boris Juelg, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (2):
  - MGH, Boston, Massachusetts
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Kenya AIDS Vaccine Initiative, Nairobi, Kenya

REFERENCES:
- See also: Related Info — http://iavi.org